CLINICAL TRIAL: NCT06809673
Title: PA.RI.GE. Study. The Prognostic Role of Inflammatory Circulating Biomarkers in HNSCC: a Prospective Multicentric Trial
Status: Enrolling by invitation | Type: Observational
Sponsor: Ospedale Policlinico San Martino (Other)
Responsible Party: Principal Investigator, Filippo Marchi, Dr, Ospedale Policlinico San Martino
Other Study IDs: PA.RI.GE.
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — complete blood count, kidney function (creatinine and glomerular filtrate), liver function (AST/GOT, ALT/GPT, total bilirubin), lactate dehydrogenase, albumin, fibrinogen, c reactive protein. Kidney and liver function sampling will be collected only before surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: blood sampling — blood sampling at baseline, 1,3,6 months after surgery and eventually when recurrence is detected.
  If adjuvant treatment is planned, blood sampling at baseline, 1 month after surgery, 1,3,6 months after the last fraction of RT and eventually when recurrence is detected.

SUMMARY:
This is a clinical, observational, non-pharmacological, multicenter, prospective case-control no-profit study to assess the prognostic role of several circulating inflammatory biomarkers

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years;
2. Written informed consent;
3. Squamous carcinoma of the hypopharynx, larynx and oral cavity;
4. Clinical stage I-IVa according to the VIII edition of AJCC staging system
5. Primary surgery as first line curative intent treatment, followed by ± adjuvant radiotherapy± chemotherapy based on the pathological findings following the NCCN guidelines

Exclusion Criteria:

1. Relapsing or metastatic disease
2. Locally advanced disease not amenable to curative intent treatment
3. Previous local or systemic treatment for head and neck cancer
4. Previous malignancies (exluding non-melanoma skin cancers) unless complete remission has been achieved at least 5 years before entering the study
5. Psychiatric disorder or known substance abuse
6. Concomitant immunosuppressive treatment
7. Concomitant immunostimulant treatment
8. Chronic inflammatory disease
9. Autoimmune disease
10. Major surgery in the previous year
11. History of recent onset of any condition which, in the investigator's opinion, could interfere with patient adherence for the entire duration of the protocol.
12. Positive serum pregnancy test for women of childbearing age. Women of childbearing potential (WOCBP) is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) and is not postmenopausal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by HNSCC (larynx, oral cavity, hypopharynx) treated with primary surgery +/- adjuvant treatment.
  Not included patient with prior tumors or other immunosuppressive/immunostimalnt treatment or disease.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
To identify a profile of circulating biomarkers in patients affected by HNSCC | 72 months
To identify a subset of patients in which biomarkers modifications might anticipate disease recurrence | 72 months

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Martino, Genoa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zahorec R. Neutrophil-to-lymphocyte ratio, past, present and future perspectives. Bratisl Lek Listy. 2021;122(7):474-488. doi: 10.4149/BLL_2021_078. PMID 34161115